CLINICAL TRIAL: NCT05135091
Title: A Study of Inhibitory Interneurons (NRTX-1001) in Drug-Resistant Unilateral Mesial Temporal Lobe Epilepsy (MTLE)
Brief Title: Study of NRTX-1001 Neural Cell Therapy in Drug-Resistant Unilateral Mesial Temporal Lobe Epilepsy (EPIC (EPIlepsy Cell Therapy))
Acronym: EPIC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Neurona Therapeutics (Industry)
Collaborators: California Institute for Regenerative Medicine (CIRM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NTE001
Record Dates: First submitted 2021-11-16; First posted 2021-11-26 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Mesial Temporal Lobe Epilepsy
Keywords: Epilepsy; MTLE; seizure; EPIC; focal seizures; hippocampus
MeSH Terms: conditions — Epilepsy; Seizures

STUDY DESIGN:
Intervention Model Description: This is a two-phase study. Phase 1/2 is an open-label, single arm, sequential dose escalation. Phase 3 is a multicenter, double-blind, randomized, parallel group, sham controlled study.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This is a two-phase study. Phase 1/2 is open-label and unmasked. Phase 3 is blinded with participant, part of investigator team, and outcomes assessor masked to treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- NRTX-1001 (Phase 1/2) (Experimental): Up to 28 subjects
  Interventions: Biological: NRTX-1001
- NRTX-1001 (Phase 3) (Experimental): Approximately 40 subjects
  Interventions: Biological: NRTX-1001
- Sham Comparator (Phase 3) (Sham Comparator): Approximately 20 subjects
  Interventions: Procedure: Sham Comparator

INTERVENTIONS:
Biological: NRTX-1001 — Biological: NRTX-1001 is an experimental neural cell therapy product candidate derived from an allogeneic human embryonic stem cell line. The stem cells were converted into inhibitory nerve cells that produce GABA.
  Other Names: GABA-secreting interneurons
  Arms: NRTX-1001 (Phase 1/2)
Biological: NRTX-1001 — Biological: NRTX-1001 is an experimental neural cell therapy product candidate derived from an allogeneic human embryonic stem cell line. The stem cells were converted into inhibitory nerve cells that produce GABA.
  Other Names: GABA-secreting interneurons
  Arms: NRTX-1001 (Phase 3)
Procedure: Sham Comparator — Sham Comparator
  Arms: Sham Comparator (Phase 3)

SUMMARY:
This clinical trial is designed to test whether a single image-guided intracerebral administration of inhibitory nerve cells, called interneurons (NRTX-1001), into subjects with drug-resistant unilateral mesial temporal lobe epilepsy (MTLE), with or without mesial temporal sclerosis (MTS), is safe (frequency of adverse events) and effective (seizure frequency). NRTX-1001 comprises human interneurons that secrete a neurotransmitter, gamma-aminobutyric acid (GABA).

DETAILED DESCRIPTION:
Subjects will undergo a single CT or MRI-guided intracerebral administration of human interneurons that secrete the inhibitory neurotransmitter, gamma-aminobutyric acid (GABA), into the temporal lobe region of the brain where the seizures are thought to arise. NRTX-1001 is intended to suppress the onset and spread of seizures. Safety, efficacy, tolerability, and effects on reducing seizure frequency and epilepsy disease symptoms will be assessed at regular intervals for 2 years after the administration of NRTX-1001. After the two-year period, subjects will be followed with quarterly phone calls and annual visits in years 3 through 5, and then annual visits in years 6 through 15. Subjects will be placed on an immunosuppressant medication regimen for a duration of one year to partially suppress the subjects' immune system to promote the intended long-term persistence of NRTX-1001. This immunosuppressant medication is intended to be discontinued after the first year; however, the NRTX-1001 cells are intended to persist long-term.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or Female, age ≥18 to ≤75
2. Focal seizures, clinically defined as unilateral MTLE
3. Has failed to achieve seizure control despite adequate trials of at least 2 ASDs at appropriate doses
4. Currently on stable doses (at least 1 month prior to Screening) of approved ASDs
5. Single seizure focus confirmed within one hippocampus
6. Seizure frequency averages ≥4 per 28-day period, including at least 2 clinical focal seizures per 28-day period with objective manifestations or more severe types, over the 6 months prior to the Screening Visit. (Phase 1/2 only)
7. Disabling seizure frequency of ≥2 per 28-day period averaged over 3 months prior to the Screening visit and over a prospective 10-week baseline period prior to Randomization (Phase 3 Only)

Key Exclusion Criteria:

1. Epilepsy due to other medical conditions and/or progressive neurologic disease
2. Evidence of seizure focus outside of the hippocampus or evidence of seizures of non- focal origin.
3. Significant other medical conditions which would impair safe participation
4. History of status epilepticus in the 3 years prior to screening.
5. Primary or secondary immunodeficiency
6. Suicide attempts in the past year 3 years
7. Severe psychiatric disorders
8. Prior lobectomy or LITT procedure
9. MRI indicating potential malignant lesion
10. Pregnancy, or currently breastfeeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2022-06-16 (Actual); Primary Completion 2029-02 (Estimated); Study Completion 2043-09 (Estimated)

PRIMARY OUTCOMES:
Frequency of serious or severe AEs (Phase 1/2) | 1 year
  The primary endpoint of the study is the frequency of serious or severe AEs over the period of 1 year after administration.
Change in disabling seizure frequency (Phase 3) | 4-6 months after surgery
  The difference in median percent change from baseline in diary-reported disabling seizure frequency (seizures per 28 days) between subjects that receive NRTX-1001 and those who receive sham treatment.

SECONDARY OUTCOMES:
Responder rate (Phase 3) | 4-6 months after surgery
  The difference in the 50% responder rate, e.g., the difference between the fraction of subjects who receive NRTX-1001 and those that receive sham treatment who experience at least a 50% reduction from baseline in disabling seizure frequency.
Responder rate (Phase 3) | 4-6 months after surgery
  The difference in the 75% responder rate, e.g., the difference between the fraction of subjects who receive NRTX-1001 and those that receive sham treatment who experience at least a 75% reduction from baseline in disabling seizure frequency.

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Dunayevich, MD, Study Director — Neurona Therapeutics
Locations (31):
- United States (31):
  - Mayo Clinic Arizona Epilepsy Center, Phoenix, Arizona
  - Banner-University of Arizona Medical Center Tucson Comprehensive Epilepsy Program, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - University of Southern California Keck Hospital, Los Angeles, California
  - University of California Los Angeles, Los Angeles, California
  - UC Irvine Medical Center, Orange, California
  - Stanford University, Palo Alto, California
  - University of California Davis, Sacramento, California
  - University of California San Diego, San Diego, California
  - University of California San Francisco, San Francisco, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - George Washington University, Washington D.C., District of Columbia
  - University of Miami, Miami, Florida
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - University of Iowa Health Care, Iowa City, Iowa
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Wayne State University/Detroit Medical Center Comprehensive Epilepsy Program, Detroit, Michigan
  - NYU Langone Comprehensive Epilepsy Center, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Atrium Health, Charlotte, North Carolina
  - Duke University Hospital, Durham, North Carolina
  - Atrium Wake Forest Baptist, Winston-Salem, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas
  - UTHealth Houston, Houston, Texas
  - University of Utah Health, Salt Lake City, Utah
  - University of Washington Regional Epilepsy Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bershteyn M, Broer S, Parekh M, Maury Y, Havlicek S, Kriks S, Fuentealba L, Lee S, Zhou R, Subramanyam G, Sezan M, Sevilla ES, Blankenberger W, Spatazza J, Zhou L, Nethercott H, Traver D, Hampel P, Kim H, Watson M, Salter N, Nesterova A, Au W, Kriegstein A, Alvarez-Buylla A, Rubenstein J, Banik G, Bulfone A, Priest C, Nicholas CR. Human pallial MGE-type GABAergic interneuron cell therapy for chronic focal epilepsy. Cell Stem Cell. 2023 Oct 5;30(10):1331-1350.e11. doi: 10.1016/j.stem.2023.08.013. PMID 37802038
- See also: Related Info — http://www.neuronatherapeutics.com